CLINICAL TRIAL: NCT02551887
Title: HPV Vaccination: An Investigation of Physician Reminders and Recommendation Scripts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenstrief Institute, Inc. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Merck - 14
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Human Papilloma Virus Infection Type 11; Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Human Papilloma Virus Infection Type 6; Cervical Cancer; Genital Warts; Oropharyngeal Cancer
Keywords: HPV Vaccinations; Quadrivalent Vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata; Oropharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Usual Care Only
- Automated Reminder (Active Comparator): Reminder
  Interventions: Behavioral: Automated Reminder
- Automated Reminder Plus Script (Experimental): Provider sees both reminder and script.
  Interventions: Behavioral: Automated Reminder Plus Script

INTERVENTIONS:
Behavioral: Automated Reminder — Automated reminder shown to provider
  Arms: Automated Reminder
Behavioral: Automated Reminder Plus Script — Provider sees both reminder and script.
  Arms: Automated Reminder Plus Script

SUMMARY:
Primary, Secondary, and Exploratory Objective(s):

Primary objective: To evaluate the effect of interventions on 1st dose uptake of HPV vaccine.

DETAILED DESCRIPTION:
Study Rationale:

Human papillomavirus (HPV) vaccine uptake among females and males remains unacceptably low. Health care provider recommendation of HPV vaccine is a major driver of vaccine acceptance. Conversely, the failure of health care providers to recommend HPV vaccine has repeatedly been identified as the primary factor in non-vaccination. Among many recommendations for increasing HPV vaccination rates are several that specifically target health care providers. Two approaches are implementation of electronic health records-based decision support systems and interventions designed to help physicians recommend HPV vaccine in a routine, matter-of-fact manner that addresses uneasiness in discussing sexual activity with parents of adolescents.

A randomized, 3-arm interventional study is proposed.

The 3 arms (randomized at the level of health care provider) will be:

1. usual practice;
2. automated reminders to recommend HPV vaccine for eligible male and female adolescents during clinic visits;
3. automated reminders PLUS a suggested recommendation script.

Here is a draft of the recommendation script that the study team is proposing for the third arm of the study: "Three vaccines are recommended for <first name>, meningococcal to prevent meningitis, HPV to prevent cancer, and Tdap to prevent tetanus. All three are recommended at this age". The script draft was based on the principles of Diffusion Theory and on theories of learning and memory.

Diffusion Theory predicts that adoption of an innovation (in this case the recommendation script) is predicted by three central factors:

1. The innovation should be seen as superior to the approach it is intended to replace (ADVANTAGE);
2. The innovation should be viewed as consistent with pre-existing beliefs and experiences (COMPATIBILITY); and
3. The innovation should be seen as easy to understand and implement (COMPLEXITY).

It is believed that the proposed script meets the ADVANTAGE criterion in that it provides a simple, straightforward way of introducing the HPV vaccine into conversations with adolescents and their parents, an issue with which some physicians struggle. The script meets the COMPATIBILITY criterion in that it makes the HPV vaccine recommendation consistent with the way other vaccines are typically recommended in conversations with adolescents and their parents. Finally, the proposed script meets the COMPLEXITY criterion in that it is simple and will likely be time-saving in most cases. Furthermore, the existing electronic health record (EHR) infrastructure at the target clinics will support easy introduction of the recommendation and script into clinical workflow.

Research in learning and memory has shown that information presented first or last in a sequence has the greatest salience and is therefore most likely to be remembered. In our suggested script, HPV vaccine was purposely in the middle, between Tdap and meningococcal vaccines to decrease the salience of HPV vaccination, thereby helping physicians to treat the three vaccines in a consistent manner. When HPV vaccine is mentioned last, there may be a tendency to hesitate or to treat it as separate from the other recommended vaccines.

Approximately 30 pediatric health care providers will be randomized across the 3 arms in equal numbers. The primary outcome of interest, HPV vaccination, will be evaluated as a patient outcome nested within provider. Physician acceptance of the recommendations, comparing changes in vaccination rates with qualitative feedback from providers will be further assessed. To gather qualitative feedback, 3-4 pediatric health care providers in each clinic will be interviewed. Participants will be purposely selected based on provider demographics, including gender, years in practice, and role within the clinic organizational structure. The interviews will be guided by the Consolidated Framework for Implementation Research (CFIR), a theory and evidence-based framework that represents the accumulated results of over 50 years of research on implementation and diffusion. Mixed methods will enable the team to examine not only impact on vaccination rates but also the characteristics of the reminder (e.g., usability, support of workflow), its implementation, and the context of setting in which it was implemented (e.g., clinical structure).

Aims and Objectives Aim 1. To evaluate the effects of physician-targeted automated HPV vaccination reminders alone and reminders plus a recommended script on HPV vaccination rates among 9-12 year old male and female patients.

Hypothesis. It is expected that a linear increase in HPV vaccination rates across the usual practice control group and the two intervention conditions, such that the reminder + script group will have the highest first dose HPV vaccination rates, followed by the reminder-only group will be noted.

Secondary objective: To evaluate rates of return for second dose. Exploratory objective: To evaluate experiences of pediatric health care providers with the reminder and script interventions.

Materials and Methods:

The Child Health Improvement through Computer Automation (CHICA) system, described in detail above, has already been developed and has been in operation since November of 2004. The functionality is well documented. New components of the system will have to be developed for this study. The first of these will be the activation of CHICA's ability to randomize its alerts by provider. The second will be the development of the Arden Syntax rules (Medical Logic Modules) to query the data from the immunization registry and generate appropriate prompts and reminders to the clinician. Once written, these rules must be encoded in CHICA and extensively tested with clinical data before they are deployed. Third, the study team will develop a mechanism by which CHICA can query the immunization registry at some time point after the clinic visit to determine whether an HPV vaccine was administered.

Include potential difficulties and limitations of the available methods and strategies for overcoming those methods. Randomization by physician depends on having accurate data from the clinic's registration system about which physician the patient will see. The study team has used this information in the past without significant problems. However, if it is noted that the data are missing or unreliable in a significant number of cases, the study team can ask for the information to be entered into the system by clinic personnel prior to the visit.

Programming of Arden rules is part and parcel of operating the CHICA system. So the study team does not anticipate problems with developing and testing these. The study team closely monitor the display and response to CHICA reminders. If there is a problem, the study team will be able to detect and correct it quickly.

The ability to query the CHIRP immunization registry by Health Level Seven International (HL7) messaging has recently been developed. The responses from CHIRP are not perfect, but are well over 90% reliable. The study team will build our system for querying CHIRP for HPV data to track and reissue failed queries in order to maximize the available data.

The location of the study sites. As previously noted, the study will be conducted in the five clinics in the Eskenazi Health System that currently use CHICA. They are: Eskenazi Outpatient Care Center, Blackburn, Pecar, Eskenazi 38th St., and Forest Manor.

Outcome measurement. The outcome of primary interest, HPV vaccine uptake, will be recorded by having the CHICA system re-query the CHIRP system after each visit. The study team will record whether HPV vaccine was administered. The CHICA system will be programmed to track patients who are enrolled in the study. Between 7 and 30 days after the clinic visit, CHICA will send an HL7 query for vaccination (VXQ) message for each patient to the CHIRP immunization registry of the Indiana State Department of Health. In response to this query message, CHIRP will send an HL7 vaccination record response (VXR) message with the patient's immunization record. Because all of the CHICA clinics report their immunization data to CHIRP, this will be a reliable way to assess whether the patient received an HPV vaccine.

Predictors of HPV vaccine uptake. The study team will use the re-query of CHIRP to determine which other vaccines (e.g., meningococcal; Tdap; influenza) were administered. Other variables of interest that will be recorded will be provider seen, patient age, and patient gender.

The 5 CHICA clinic study sites are located throughout metropolitan Indianapolis. These clinics serve largely low income (70% Medicaid) and minority (33% Hispanic, 49% African American) children. CHICA has provided data to over 37,000 children since first implemented in 2004. As indicated in Part 1 (Introduction), these CHICA clinics have been used successfully for multiple pediatric health service intervention studies. The real-world implementation being used in this study is a great strength. It will enable us to evaluate how a reminder system and recommended script influence HPV vaccination practices in busy pediatric clinics. An inherent limitation with this kind of study is that the study team is limited in the kind of data that can be collected. The study team cannot, for instance, collect attitude/knowledge information from parents. However, it is believed that the strengths of this research methodology far outweigh the limitations.

Qualitative interviews. Interviews will be digitally recorded and transcribed. Interviewers will be asked to record field notes related to the interview to capture information not included in the transcripts (e.g., tone of voice). Digital recordings will be transferred to a password-protected computer, in a locked office. Recordings and transcripts will be saved for a 3-year period from the end of the study. At that point in time, digital recordings and transcripts will be permanently erased. Content analysis will enable investigators to identify patterns in respondents' answers. The study team will specifically look for barriers to implementation and use of the recommendations and scripts as well as contextual aspects that facilitated routine use of the recommendations and scripts to improve adherence to recommended HPV vaccination guidelines.

ELIGIBILITY:
Inclusion Criteria:

Eligible Providers

* All pediatricians and nurse practitioners who provide health care at the 5 CHICA clinics will be included in this study.

Eligible Patients

* Males and females
* 11-14 years of age with no prior HPV vaccine doses administered
* Eligible for Tdap and/or MCV4 vaccination at the visit.

Exclusion Criteria:

* Patients in the eligible age range who have already received one or more of the adolescent platform vaccines

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 647 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parkin DM, Bray F. Chapter 2: The burden of HPV-related cancers. Vaccine. 2006 Aug 31;24 Suppl 3:S3/11-25. doi: 10.1016/j.vaccine.2006.05.111. PMID 16949997
- [Background] Giuliano AR, Anic G, Nyitray AG. Epidemiology and pathology of HPV disease in males. Gynecol Oncol. 2010 May;117(2 Suppl):S15-9. doi: 10.1016/j.ygyno.2010.01.026. Epub 2010 Feb 6. PMID 20138345
- [Background] Chaturvedi AK. Beyond cervical cancer: burden of other HPV-related cancers among men and women. J Adolesc Health. 2010 Apr;46(4 Suppl):S20-6. doi: 10.1016/j.jadohealth.2010.01.016. PMID 20307840
- [Background] Haupt RM, Sings HL. The efficacy and safety of the quadrivalent human papillomavirus 6/11/16/18 vaccine gardasil. J Adolesc Health. 2011 Nov;49(5):467-75. doi: 10.1016/j.jadohealth.2011.07.003. Epub 2011 Sep 9. PMID 22018560
- [Background] Global Advisory Committee on Vaccine Safety,12-13 June 2013. Wkly Epidemiol Rec. 2013 Jul 19;88(29):301-12. No abstract available. English, French. PMID 23909011
- [Background] Arnheim-Dahlstrom L, Pasternak B, Svanstrom H, Sparen P, Hviid A. Autoimmune, neurological, and venous thromboembolic adverse events after immunisation of adolescent girls with quadrivalent human papillomavirus vaccine in Denmark and Sweden: cohort study. BMJ. 2013 Oct 9;347:f5906. doi: 10.1136/bmj.f5906. PMID 24108159
- [Background] Ojha RP, Jackson BE, Tota JE, Offutt-Powell TN, Singh KP, Bae S. Guillain-Barre syndrome following quadrivalent human papillomavirus vaccination among vaccine-eligible individuals in the United States. Hum Vaccin Immunother. 2014;10(1):232-7. doi: 10.4161/hv.26292. Epub 2013 Sep 6. PMID 24013368
- [Background] Klein NP, Hansen J, Chao C, Velicer C, Emery M, Slezak J, Lewis N, Deosaransingh K, Sy L, Ackerson B, Cheetham TC, Liaw KL, Takhar H, Jacobsen SJ. Safety of quadrivalent human papillomavirus vaccine administered routinely to females. Arch Pediatr Adolesc Med. 2012 Dec;166(12):1140-8. doi: 10.1001/archpediatrics.2012.1451. PMID 23027469
- [Background] Pedersen C, Petaja T, Strauss G, Rumke HC, Poder A, Richardus JH, Spiessens B, Descamps D, Hardt K, Lehtinen M, Dubin G; HPV Vaccine Adolescent Study Investigators Network. Immunization of early adolescent females with human papillomavirus type 16 and 18 L1 virus-like particle vaccine containing AS04 adjuvant. J Adolesc Health. 2007 Jun;40(6):564-71. doi: 10.1016/j.jadohealth.2007.02.015. PMID 17531764
- [Background] Reisinger KS, Block SL, Lazcano-Ponce E, Samakoses R, Esser MT, Erick J, Puchalski D, Giacoletti KE, Sings HL, Lukac S, Alvarez FB, Barr E. Safety and persistent immunogenicity of a quadrivalent human papillomavirus types 6, 11, 16, 18 L1 virus-like particle vaccine in preadolescents and adolescents: a randomized controlled trial. Pediatr Infect Dis J. 2007 Mar;26(3):201-9. doi: 10.1097/01.inf.0000253970.29190.5a. PMID 17484215
- [Background] Baandrup L, Blomberg M, Dehlendorff C, Sand C, Andersen KK, Kjaer SK. Significant decrease in the incidence of genital warts in young Danish women after implementation of a national human papillomavirus vaccination program. Sex Transm Dis. 2013 Feb;40(2):130-5. doi: 10.1097/OLQ.0b013e31827bd66b. PMID 23324976
- [Background] Ali H, Donovan B, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Guy RJ. Genital warts in young Australians five years into national human papillomavirus vaccination programme: national surveillance data. BMJ. 2013 Apr 18;346:f2032. doi: 10.1136/bmj.f2032. PMID 23599298
- [Background] Ali H, Guy RJ, Wand H, Read TR, Regan DG, Grulich AE, Fairley CK, Donovan B. Decline in in-patient treatments of genital warts among young Australians following the national HPV vaccination program. BMC Infect Dis. 2013 Mar 18;13:140. doi: 10.1186/1471-2334-13-140. PMID 23506489
- [Background] Centers for Disease Control and Prevention (CDC). National and state vaccination coverage among adolescents aged 13-17 years--United States, 2012. MMWR Morb Mortal Wkly Rep. 2013 Aug 30;62(34):685-93. PMID 23985496
- [Background] Brewer NT, Gottlieb SL, Reiter PL, McRee AL, Liddon N, Markowitz L, Smith JS. Longitudinal predictors of human papillomavirus vaccine initiation among adolescent girls in a high-risk geographic area. Sex Transm Dis. 2011 Mar;38(3):197-204. doi: 10.1097/OLQ.0b013e3181f12dbf. PMID 20838362
- [Background] Guerry SL, De Rosa CJ, Markowitz LE, Walker S, Liddon N, Kerndt PR, Gottlieb SL. Human papillomavirus vaccine initiation among adolescent girls in high-risk communities. Vaccine. 2011 Mar 9;29(12):2235-41. doi: 10.1016/j.vaccine.2011.01.052. Epub 2011 Feb 1. PMID 21288799
- [Background] Liddon NC, Hood JE, Leichliter JS. Intent to receive HPV vaccine and reasons for not vaccinating among unvaccinated adolescent and young women: findings from the 2006-2008 National Survey of Family Growth. Vaccine. 2012 Mar 30;30(16):2676-82. doi: 10.1016/j.vaccine.2012.02.007. Epub 2012 Feb 15. PMID 22342548
- [Background] Zimet GD, Weiss TW, Rosenthal SL, Good MB, Vichnin MD. Reasons for non-vaccination against HPV and future vaccination intentions among 19-26 year-old women. BMC Womens Health. 2010 Sep 1;10:27. doi: 10.1186/1472-6874-10-27. PMID 20809965
- [Background] Vadaparampil ST, Kahn JA, Salmon D, Lee JH, Quinn GP, Roetzheim R, Bruder K, Malo TL, Proveaux T, Zhao X, Halsey N, Giuliano AR. Missed clinical opportunities: provider recommendations for HPV vaccination for 11-12 year old girls are limited. Vaccine. 2011 Nov 3;29(47):8634-41. doi: 10.1016/j.vaccine.2011.09.006. Epub 2011 Sep 14. PMID 21924315
- [Background] Evans, G. and A. Bostrom, The evolution of vaccine risk communication in the United States: 1982-2002, in Jordan report 20th anniversary: Accelerated development of vaccines 2002, A. National Institute of and D. Infectious, Editors. 2002, U.S. Department of Health and Human Services, National Institute of Allergy and Infectious Diseases: Washington, D.C. p. 58-71.
- [Background] Esposito S, Bosis S, Pelucchi C, Begliatti E, Rognoni A, Bellasio M, Tel F, Consolo S, Principi N. Pediatrician knowledge and attitudes regarding human papillomavirus disease and its prevention. Vaccine. 2007 Aug 29;25(35):6437-46. doi: 10.1016/j.vaccine.2007.06.053. Epub 2007 Jul 16. PMID 17673339
- [Background] Schnatz PF, Humphrey K, O'Sullivan DM. Assessment of the perceptions and administration of the human papillomavirus vaccine. J Low Genit Tract Dis. 2010 Apr;14(2):103-7. doi: 10.1097/LGT.0b013e3181b240ca. PMID 20354417
- [Background] Kahn JA. Vaccination as a prevention strategy for human papillomavirus-related diseases. J Adolesc Health. 2005 Dec;37(6 Suppl):S10-6. doi: 10.1016/j.jadohealth.2005.08.018. PMID 16310136
- [Background] Ko EM, Missmer S, Johnson NR. Physician attitudes and practice toward human papillomavirus vaccination. J Low Genit Tract Dis. 2010 Oct;14(4):339-45. doi: 10.1097/LGT.0b013e3181dca59c. PMID 20885162
- [Background] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for ADHD diagnosis: a randomized controlled trial. Pediatrics. 2013 Sep;132(3):e623-9. doi: 10.1542/peds.2013-0933. Epub 2013 Aug 19. PMID 23958768
- [Background] Carroll AE, Biondich P, Anand V, Dugan TM, Downs SM. A randomized controlled trial of screening for maternal depression with a clinical decision support system. J Am Med Inform Assoc. 2013 Mar-Apr;20(2):311-6. doi: 10.1136/amiajnl-2011-000682. Epub 2012 Jun 28. PMID 22744960
- [Background] Carroll AE, Biondich PG, Anand V, Dugan TM, Sheley ME, Xu SZ, Downs SM. Targeted screening for pediatric conditions with the CHICA system. J Am Med Inform Assoc. 2011 Jul-Aug;18(4):485-90. doi: 10.1136/amiajnl-2011-000088. PMID 21672910
- [Background] Fiks AG, Grundmeier RW, Mayne S, Song L, Feemster K, Karavite D, Hughes CC, Massey J, Keren R, Bell LM, Wasserman R, Localio AR. Effectiveness of decision support for families, clinicians, or both on HPV vaccine receipt. Pediatrics. 2013 Jun;131(6):1114-24. doi: 10.1542/peds.2012-3122. Epub 2013 May 6. PMID 23650297
- [Background] Markowitz LE, Hariri S, Lin C, Dunne EF, Steinau M, McQuillan G, Unger ER. Reduction in human papillomavirus (HPV) prevalence among young women following HPV vaccine introduction in the United States, National Health and Nutrition Examination Surveys, 2003-2010. J Infect Dis. 2013 Aug 1;208(3):385-93. doi: 10.1093/infdis/jit192. Epub 2013 Jun 19. PMID 23785124
- [Background] Zimet GD, Rosberger Z, Fisher WA, Perez S, Stupiansky NW. Beliefs, behaviors and HPV vaccine: correcting the myths and the misinformation. Prev Med. 2013 Nov;57(5):414-8. doi: 10.1016/j.ypmed.2013.05.013. Epub 2013 May 31. PMID 23732252
- [Background] Rogers EM. A prospective and retrospective look at the diffusion model. J Health Commun. 2004;9 Suppl 1:13-9. doi: 10.1080/10810730490271449. PMID 14960401
- [Background] Glanzer, M. and A.R. Cunitz, Two storage mechanisms in free recall. Journal of Verbal Learning and Verbal Behavior, 1966. 5(4): p. 351-360.
- [Background] Rogers, E.M., Diffusion of innovations. Vol. 4th 1995, New York: Free Press.
- [Background] Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. Milbank Q. 2004;82(4):581-629. doi: 10.1111/j.0887-378X.2004.00325.x. PMID 15595944
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Anand V, Biondich PG, Liu G, Rosenman M, Downs SM. Child Health Improvement through Computer Automation: the CHICA system. Stud Health Technol Inform. 2004;107(Pt 1):187-91. PMID 15360800
- [Background] Anand V, Carroll AE, Downs SM. Automated primary care screening in pediatric waiting rooms. Pediatrics. 2012 May;129(5):e1275-81. doi: 10.1542/peds.2011-2875. Epub 2012 Apr 16. PMID 22508925
- [Background] Biondich PG, Downs SM, Anand V, Carroll AE. Automating the recognition and prioritization of needed preventive services: early results from the CHICA system. AMIA Annu Symp Proc. 2005;2005:51-5. PMID 16779000
- [Background] Downs SM, Uner H. Expected value prioritization of prompts and reminders. Proc AMIA Symp. 2002:215-9. PMID 12463818
- [Background] Downs SM, Zhu V, Anand V, Biondich PG, Carroll AE. The CHICA smoking cessation system. AMIA Annu Symp Proc. 2008 Nov 6;2008:166-70. PMID 18998823
- [Background] Bauer, N.S., et al., Computer Decision Support to Improve Autism Screening and Care in Community Pediatric Clinics. Infants & Young Children, 2013. 26(4): p. 306-317.
- [Background] Denzin, N.K. and Y.S. Lincoln, The Sage handbook of qualitative research. Vol. 4th. 2011, Thousand Oaks, CA: Sage.
- [Background] Braun, V. and V. Clarke, Using thematic analysis in psychology. Qualitative research in psychology, 2006. 3(2): p. 77-101.
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475
- [Derived] Dixon BE, Kasting ML, Wilson S, Kulkarni A, Zimet GD, Downs SM. Health care providers' perceptions of use and influence of clinical decision support reminders: qualitative study following a randomized trial to improve HPV vaccination rates. BMC Med Inform Decis Mak. 2017 Aug 10;17(1):119. doi: 10.1186/s12911-017-0521-6. PMID 28797293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 15, 2014 - April 30, 2015
  Locations: The 5 CHICA clinic study sites were located throughout metropolitan Indianapolis. These clinics serve largely low income (70% Medicaid) and minority (33% Hispanic, 49% African American) children. CHICA has provided data to over 37,000 children since first implemented in 2004.
Groups:
- Usual Care: Non-interventional study arm. Patients receive usual care.
- Automated Reminder: Automated Reminder: Health care providers were given a list of vaccines to consider for administration (MCV4; HPV; Tdap) and asked to check the shots given.
- Automated Reminder Plus Recommended Script: Automated Reminder Plus Recommended Script: In addition to the list of vaccines, health care providers were given a suggested script for recommending vaccination.
Period: Overall Study
Arm/Group | Usual Care | Automated Reminder | Automated Reminder Plus Recommended Script
Started | 301 | 124 | 222
Completed | 301 | 124 | 222
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: These were eligible patients males and females 11-14 years of age with no prior HPV vaccine doses administered. Additionally, they also had to be eligible for Tdap and/or MCV4 vaccination at the visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Automated Reminder | Automated Reminder Plus Recommended Script | Total
Number analyzed (Participants) | 301 | 124 | 222 | 647
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 301 | 124 | 222 | 647
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 56 | 105 | 291
  Male | 171 | 68 | 117 | 356
Region of Enrollment [Number; unit: Participants]
  United States | 301 | 124 | 222 | 647

OUTCOME MEASURES:

1. Primary Outcome: First Dose HPV Vaccine Uptake
Description: The outcome of primary interest, HPV vaccine uptake, is recorded as the number of patients who receive the first dose of HPV vaccine.
Time Frame: Nine Months
Population: Number of patients that received the first dose of HPV vaccine.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Automated Reminder | Automated Reminder Plus Recommended Script
Number analyzed (Participants) | 301 | 124 | 222
Participants | 118 | 63 | 117

2. Secondary Outcome: Second Dose HPV Vaccine Uptake
Description: The rate of second dose of HPV vaccine uptake, is recorded as the number of patients who receive the second dose of HPV vaccine.
Time Frame: Nine Months
Population: Number in the control condition who were eligible for 2 doses of vaccine.
Measure: Number; unit: Participants
Arm/Group | Usual Care | Automated Reminder | Automated Reminder Plus Recommended Script
Number analyzed (Participants) | 235 | 97 | 172
Participants | 20 | 8 | 17

ADVERSE EVENTS:
Time Frame: 10 Months
Description: Data was collected for ten months, and no adverse event occurred.
Groups:
- Usual Care: Patients receive usual care.
- Automated Reminder: Health care providers were given a list of vaccines to consider for administration (MCV4; HPV; Tdap) and asked to check the shots given.
- Automated Reminder Plus Recommended Script: In addition to the list of vaccines, health care providers were given a suggested script for recommending vaccination.
Arm/Group | Usual Care | Automated Reminder | Automated Reminder Plus Recommended Script
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/124 | 0/222
Other Adverse Events (participants affected / at risk) | 0/301 | 0/134 | 0/222

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No